CLINICAL TRIAL: NCT04774562
Title: The Effect of Video-Assisted Discharge Education After Total Hip Replacement Surgery on Activities of Daily Living, Functionality and Patient Satisfaction: A Randomized Controlled Study
Brief Title: The Effect of Video-Assisted Discharge Education After Total Hip Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ozum Cetinkaya Eren (Other)
Collaborators: Pamukkale University (Other); Akdeniz University (Other)
Responsible Party: Sponsor-Investigator, Ozum Cetinkaya Eren, Academician, Alanya Alaaddin Keykubat University
Organization: Alanya Alaaddin Keykubat University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VADEafterTHR
Record Dates: First submitted 2021-02-20; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Total Hip Replacement; Patient Education; Patient Satisfaction; Activities of Daily Living
Keywords: Patient education; Function; Kinesiophobia; Total Hip Replacement
MeSH Terms: conditions — Patient Satisfaction; Kinesiophobia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This study included 31 participants who were randomly divided in the physiotherapy (PT) group (n=18), and the video-assisted discharge education (VADE) group (n=13). Both groups received a physiotherapy program. VADE group was additionally received VADE program. The physiotherapy program included breathing exercises, positioning, hip range of motion and strengthening exercises, and information about walking and ambulation. The VADE program included information about THR, preventive rehabilitation approaches, transfer activities, using stairs, self-care activities, home settings by modifying the treatment and discharge protocols of Lucas (2008). The whole program was taught verbally and practically and a physiotherapy booklet prepared with the same content was given to the participants and their relatives.
Who Masked: Participant
Masking Description: Patients and their relatives were given physiotherapy and video-assisted discharge education by the same physiotherapist without being told which group they were in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-Assisted Discharge Education (VADE) Group (Experimental): VADE group received video-assisted discharge education in addition to the physiotherapy program given to the PT group on the same day by the same physiotherapist. The VADE program included information about THR, preventive rehabilitation approaches, transfer activities, using stairs, self-care activities, home settings. VADE was prepared as a presentation of written information and videos which is shown this information by a professional model. Video shoots were done by a physiotherapist experienced in the field of physiotherapy and rehabilitation after THR surgery. The presentation was stopped when participants have questions or have points were not understood and the necessary explanations were shown verbally and practically. Along with the physiotherapy booklet, the participants were given an educational booklet containing written and visual information prepared in the same content as VADE.
  Interventions: Behavioral: Video-Assisted Discharge Education (VADE); Behavioral: Physiotherapy (PT) Program
- Physiotherapy (PT) Group (Experimental): The physiotherapy program given to the PT group after THR surgery. The physiotherapy program included breathing exercises, positioning, hip range of motion and strengthening exercises, and information about walking and ambulation. The whole program was taught verbally and practically to participants and their relatives. Information was given about the exercises to be added at the end of the first week and in the 4th week. A physiotherapy booklet prepared with the same content was given to the participants. The booklet was examined by the patient and relatives, and the questions they asked were answered by the same physiotherapist. The participants were informed that they should continue the exercises for 12 weeks.
  Interventions: Behavioral: Physiotherapy (PT) Program

INTERVENTIONS:
Behavioral: Video-Assisted Discharge Education (VADE) — Video-Assisted Discharge Education (VADE): Information about THR, preventive rehabilitation approaches, transfer activities, using stairs, self-care activities.
  Arms: Video-Assisted Discharge Education (VADE) Group
Behavioral: Physiotherapy (PT) Program — Physiotherapy (PT): Breathing exercises, positioning, hip range of motion and strengthening exercises, and information about walking and ambulation.

SUMMARY:
Abstract Objective: The aim of this study was to investigate the effect of a video-assisted discharge education program on activities of daily living, functionality, and patient satisfaction after total hip replacement (THR) surgery.

Methods: This study included 31 participants who were randomly divided in the physiotherapy (PT) group (n=18), and the video-assisted discharge education (VADE) group (n=13). Both groups received a physiotherapy program. VADE group was additionally received VADE program. In both groups, all education programs were given face to face. Data were collecting using visual analog scale (VAS), Harris Hip Score (HHS), Nottingham Extended Activities of Daily Living Scale (NEADL), Tampa Scale of Kinesiophobia (TSK) and Patient Satisfaction Questionnaire at 1st week and 3rd month.

Practice Implications: The current study has contributed to the development of video-assisted health technologies.

DETAILED DESCRIPTION:
Total Hip Replacement (THR) is a common surgical procedure performed in patients who do not respond to long-term conservative treatment to reduce high pain sensation and movement limitation in the joint (Li and Xu, 2018). Physiotherapy and rehabilitation routinely applied to regain functional independence in daily living, restore pain and joint range of motion, eliminate muscle weakness, regulate walking pattern, prevent falls, loosening, revision surgery and dislocations in the prosthesis, increase participation in activities of daily living (ADL), quality of life (QoL) and patient satisfaction levels after THR (Louw et al., 2013; Galea et al., 2008). It was determined in Kennedy et al. (2017) that patients have education expectations on recognition of the surgical team, general information about the disease and prosthesis, rehabilitation, pain management, home care activities, complications, medications, ADL after THR surgery. At the present time, with the help of demographic changes in the society and patients, changes in healthcare provision, and technological approaches, discharge education became more effective with video assistance (Abu Abed et al., 2014). The aim of our study was to investigate the effect of a video-assisted discharge education program on activities of daily living, functionality, and patient satisfaction after total hip replacement surgery.

Methods:

The study was approved by the Non-invasive Clinical Researches Ethics Committee (60116787-020/58408) on 04.09.2018. The participants included in the study were informed about the study and informed consent form was signed by all participants. Our study was performed between September 2018 and June 2019.

Of the 36 participants who met the inclusion criteria, 5 were excluded from the study for missing follow-ups or not wanting to participate in the study. The 31 participants included in the study were randomized using systematic sampling. According to last number of file numbers odd numbers included in the physiotherapy (PT) group (n=18), and even numbers included in the video-assisted discharge education (VADE) group (n=13). The first meeting with participants was made in the hospital room within the first 5 days after THR surgery in both groups. Participants and their relatives were given physiotherapy and video-assisted discharge education by the same physiotherapist without being told which group they were in.

The physiotherapy program given to the PT group included breathing exercises, positioning, hip range of motion and strengthening exercises, and information about walking and ambulation. The whole program was taught verbally and practically to participants and their relatives. Information was given about the exercises to be added at the end of the first week and in the 4th week. A physiotherapy booklet prepared with the same content was given to the participants. The booklet was examined by the patient and relatives, and the questions they asked were answered by the same physiotherapist. The participants were informed that they should continue the exercises for 12 weeks.

VADE group received video-assisted discharge education in addition to the physiotherapy program given to the PT group on the same day by the same physiotherapist. The VADE program included information about THR, preventive rehabilitation approaches, transfer activities, using stairs, self-care activities, home settings by modifying the treatment and discharge protocols of Lucas (2008). VADE was prepared as a presentation of written information and videos which is shown this information by a professional model. Video shoots were done by a physiotherapist experienced in the field of physiotherapy and rehabilitation after THR surgery. The presentation was stopped when participants have questions or have points were not understood and the necessary explanations were shown verbally and practically. Along with the physiotherapy booklet, the participants were given an educational booklet containing written and visual information prepared in the same content as VADE. The booklet was examined by the patient and relatives during VADE, and the questions they asked were answered by the same physiotherapist.

Patient interviews were completed in approximately 30 minutes in the PT group and approximately 45 minutes in the VADE group. A healthy person was used to prevent damage to the hip joints of those who had undergone surgery in photographs and videos in the VADE and booklets. In the booklets, easily understandable sentences were used by participants and their relatives. Booklets were prepared in Arial font and 11-point size. All participants were called by phone every 15 days for 12 weeks, and their participation in the exercises and ADL was followed.

Assessments were performed within the first 5 days after the THR surgery (Descriptive Information, Pain, Patient Satisfaction Questionnaire) in the hospital room after physiotherapy and VADE programs, and at the 3rd-month control (Pain, Harris Hip Score (HHS), Tampa Scale of Kinesiophobia (TSK), Nottingham Extended Activities of Daily Living Scale (NEADL), Patient Satisfaction Questionnaire) in orthopedics and traumatology clinic.

Statistical Analysis:

In the statistical analysis of data obtained in this study, Windows-based SPSS (IBM SPSS Statistics, Version 24.0, Armonk, NY, USA) package program was used. It was calculated that the number of patients included in our study was 89% power and 95% confidence for each group. Continuous variables were expressed as a mean ± standard deviation or as a median (minimum-maximum values), and categorical variables as a number and percent. Analytical (Kolmogorov-Smirnov/Shapiro-Wilks test) and visual (Histogram and probability graphs) methods were used to test the conformity of data for normal distribution. When the parametric test assumptions were provided, Independent Sample T-Test was used to compare independent group differences; when the parametric test assumptions were not provided, Mann Whitney-U test was used to compare independent group differences. In the dependent group analyzes; when the parametric test assumptions were provided, Paired Sample T-Test was used; when the parametric test assumptions were not provided, Wilcoxon Test was used. Chi-Square Analysis and Fisher Exact Test were used compare differences between categorical variables

ELIGIBILITY:
Inclusion Criteria:

* Who can understand the verbal and written information provided to the study
* Who open to communication and cooperation

Exclusion Criteria:

* Who with neurological and metabolic diseases that may cause functional impairment
* Who previously underwent prosthetic surgery from the same or opposite lower extremities,
* Who have mental and cognitive dysfunction
* Who are morbidly obese (body mass index>40 kg/m2)
* Who did not come to at least one of the post-surgical evaluations for any reason
* Who wanted to leave the study at their own request
* Who could not continue to work due to any additional discomfort developed

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Physical Function | HHS was performed at the 3rd-month control. (Assessment took 5 minutes)
  Harris Hip Score (HHS) was used to evaluate hip physical function.
Activities of Daily Living | NEADL was performed at the 3rd-month control. (Assessment took 3 minutes)
  Activities of Daily Living of the participants was evaluated with the Nottingham Extended Activities of Daily Living Scale (NEADL).
Change in Patient Satisfaction | Patient Satisfaction questionnaire was performed within the first 5 days after the THR surgery and at the 3rd-month control. (Assessment took 2 minutes)
  Patient Satisfaction questionnaire with 5 questions prepared by the researchers was used to evaluate the satisfaction levels of the participants.

SECONDARY OUTCOMES:
Change in Pain-Visual analog scale | VAS was performed within the first 5 days after the THR surgery and at the 3rd-month control. (Assessment took 2 minutes)
  Pain of patients during sleep, rest and activity were evaluated using a visual analog scale (VAS).
Kinesiophobia | TSK was performed at the 3rd-month control. (Assessment took 3 minutes)
  Kinesiophobia was evaluated with Tampa Scale of Kinesiophobia (TSK).
Descriptive Information | Descriptive information Form was performed within the first 5 days after the THR surgery. (Assessment took 3 minutes)
  Descriptive information of the patients was documented with a prepared form.

CONTACTS AND LOCATIONS:
Overall Officials: Ozum Cetinkaya Eren, PT, MSc., Principal Investigator — Alanya Alaaddin Keykubat University; Nihal Buker, Assoc.Prof., Study Director — Pamukkale University; Hasan Atacan Tonak, Asst.Prof., Study Chair — Akdeniz University; Mustafa Urguden, Prof. Dr., Study Chair — Akdeniz University
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Q, Xu B. Oral risedronate increases Gruen zone bone mineral density after primary total hip arthroplasty: a meta-analysis. J Orthop Surg Res. 2018 Jun 7;13(1):144. doi: 10.1186/s13018-018-0794-1. PMID 29880021
- [Background] Lucas B. Total hip and total knee replacement: postoperative nursing management. Br J Nurs. 2008 Dec 11-2009 Jan 7;17(22):1410-4. doi: 10.12968/bjon.2008.17.22.31866. PMID 19057500
- [Background] Galea MP, Levinger P, Lythgo N, Cimoli C, Weller R, Tully E, McMeeken J, Westh R. A targeted home- and center-based exercise program for people after total hip replacement: a randomized clinical trial. Arch Phys Med Rehabil. 2008 Aug;89(8):1442-7. doi: 10.1016/j.apmr.2007.11.058. Epub 2008 Jun 30. PMID 18586222
- [Result] Louw A, Diener I, Butler DS, Puentedura EJ. Preoperative education addressing postoperative pain in total joint arthroplasty: review of content and educational delivery methods. Physiother Theory Pract. 2013 Apr;29(3):175-94. doi: 10.3109/09593985.2012.727527. Epub 2012 Oct 4. PMID 23035767
- [Result] Kennedy D, Wainwright A, Pereira L, Robarts S, Dickson P, Christian J, Webster F. A qualitative study of patient education needs for hip and knee replacement. BMC Musculoskelet Disord. 2017 Oct 12;18(1):413. doi: 10.1186/s12891-017-1769-9. PMID 29025397
- [Result] Abu Abed M, Himmel W, Vormfelde S, Koschack J. Video-assisted patient education to modify behavior: a systematic review. Patient Educ Couns. 2014 Oct;97(1):16-22. doi: 10.1016/j.pec.2014.06.015. Epub 2014 Jul 5. PMID 25043785

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT04774562/Prot_SAP_000.pdf